CLINICAL TRIAL: NCT05357027
Title: A Phase I/II Clinical Trail of TC-E202 Targeting HPV16 E6 for Relapsed/Refractory to Standard Treatment or Metastatic Cervical Carcinoma
Brief Title: HPV16 E6 TCR T Cells for Cervical Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to strategic portfolio decision to reallocate resources to higher-priority programs
Sponsor: TCRCure Biopharma Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-E202-CC-PI
Record Dates: First submitted 2022-01-03; First posted 2022-05-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cervical Carcinoma
Keywords: HPV16 E6; TCR T Cells; Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interleukin-2; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TC-E202 dose (Experimental): This study uses the "3+3" dose escalation method. The initial dose is Dose1, the maximum dose that patients can tolerate is determined as the phase II recommended dose (RPIID), and at least 6 patients are receiving RPIID treatment . If patients develop intolerance in Dose 1 (≥3 subjects with DLT), then the subsequent enrolled patients will receive Dose-1 infusion.
  Interventions: Biological: TC-E202 cells; Drug: IL-2; Drug: Fludarabine; Drug: Cyclophosphamide Capsules

INTERVENTIONS:
Biological: TC-E202 cells — T cells genetically engineered with a TCR targeting HPV16 E6 (E6 TCR) that display specific reactivity against HLA-A2+, HPV-16+ target cells
  Other Names: TCR T Cells
Drug: IL-2 — Following cell infusion, the patient receives high-dose bolus IL-2, which is dosed to individual patient tolerance. IL-2 improves the survival of TC-E202 cells after infusion.
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: Cyclophosphamide Capsules — Part of the non-myeloablative lymphocyte-depleting preparative regimen.

SUMMARY:
Background:

Cervical cancer is the most common gynecologic malignant tumor. The occurrence and progression of cervical carcinoma is firmly relevant to HPV (Human papilloma virus) infection. Cancer cells infected by HPV expressing an HPV protein called E6. E6 is the main factors of HPV 16 carcinogenesis. In TCR-T therapy, researchers take the blood of a certain patient, select T cells and insert genes into the cell that expressing a kind of protein that targeting HPV E6. The genetically engineered cells are called E6 TCR-T cells. The engineered cells are re-infused in the patients with cervical carcinoma.

Objective:

To evaluate the safety and efficacy of TCR-T cells in the treatment of cervical carcinoma.

Eligibility:

Adults aging 18-70 with relapsed/refractory to standard treatment or metastatic cervical carcinoma.

Design:

Patients will have many screening tests, including imaging procedures, heart and lung tests, and lab tests.

Patients will have leukapheresis. Blood will be removed through a needle in the arm. A machine separates the white blood cells. The rest of the blood is returned through a needle in the other arm.

Engineered T cells will be re-infused into the patients will stay in hospital and be evaluated.

DETAILED DESCRIPTION:
Background:

Cervical cancer is the most common gynecologic malignant tumor. The occurrence and progression of cervical carcinoma is firmly relevant to HPV (Human papilloma virus) infection.

Cancer cells infected by HPV expressing an HPV protein called E6. E6 is the main factors of HPV 16 carcinogenesis. T cells genetically engineered with a TCR targeting HPV-16 E6 (E6 TCR) display specific reactivity against HLA-A2+, HPV-16+ target cells.

T cell receptor (TCR) gene engineered T cells infusion can induce objective tumor responses in certain malignancies including HPV-16+ cancer.

Objective:

Phase I: Determine the safety and tolerability of TC-E202 inHPV16 positive patients with relapsed/refractory to standard treatment or metastatic cervical carcinoma and determine the Recommended Phase II Dose (RPIID).

Primary endpoints: safety and tolerability. The evaluation of safety and tolerability will be based on the following endpoints: 1) Whether DLT occurs or MTD is achieved; 2) The incidence of various adverse events and serious adverse events and their relationship with TCR-T, IL-2, lymphodepletion chemotherapy and leukapheresis.

Secondary endpoints: efficacy. Objective response rate (ORR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS) were assessed based on RECIST 1.1 and iRECIST.

Eligibility:

Adults aging 18-70 with relapsed/refractory to standard treatment or metastatic cervical carcinoma.

Eligible patients were HLA-A*02 and had metastatic HPV16-positive cervical cancer. Patients had received or declined previous systemic therapy, with more than 4 weeks elapsed since previous systemic treatment. Patients had an Eastern Cooperative Oncology Group performance score of 0 or 1 and adequate hematologic, hepatic, and renal function.

Design:

This is a Phase I/II clinical trial to evaluate the efficacy and safety of TC-E202.

Dose escalation will proceed according to 3+3 procedure. All patients will receive a lymphocyte-depleting preparative regimen of cyclophosphamide and fludarabine followed by an infusion of E6 TCR (TC-E202) cells. Cell infusion will be followed by IL-2 administration.

All patents will be evaluated based on ORR according to RECIST v1.1&iRECIST. Phase I clinical trials establish a Drug Safety Review Committee (SRC), and the SRC will hold regular and irregular meetings to evaluate the safety data of the subjects, the clinical pharmacology, along with associated clinical efficacy, to decide escalating dose and RPIID. In addition, the SRC will decide whether to explore higher or lower doses than planned doses based on specific data.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and sign the Informed of Consent Document. Be willing to follow the procedure and protocol of the clinical trial.
2. Age ≥ 18 years and ≤ 70 years.
3. Expected survival time > 3 months.
4. ECOG score 0-1.
5. Recurrent or metastatic cervical carcinoma based on TNM & FIGO staged histopathological investigation.
6. Received at least second-line standard treatment and diagnosed as PD through image assessment. (previously received radio-therapy, chemo-therapy, targeted-therapy or immune-therapy, wash-out period > 14 or 5 half life)
7. Be able provide fresh or preserved tissue specimen. (fresh specimen first, paraffine specimen or at least 12 tumor section, tumor tissue >20%)
8. At least 1 measurable lesion (according to RECIST1.1 standard）.
9. HPV16 positive.
10. HLA-A2 positive.
11. Hematology should at least meet the following criteria:

    Absolute neutrophil count (ANC) ≥ 1.5× 109/L (±20%)； Platelet (PLT） ≥ 75× 109/L (±20%）； Hemoglobin (HGB) ≥ 90 g/L (±20%).
12. Blood biochemistry should at least meet the following criteria:

    Serum creatinine (Cr) ≤ 1.5 times of upper limit of normal (ULN) or creatine clearance ≥ 60 ml/min; Serum Alanine aminotransferase (ALT) or/and Aspartate aminotransferase (AST) ≤ 2.5 times of upper limit of normal; Total bilirubin (TBIL) ≤ 15 times of upper limit of normal.
13. Blood coagulation function is normal: Prothrombin time (PT) ≤ 1.5 ULN, International Normalized Ratio (INR) ≤ 1.5 ULN, or Activated Partial Thromboplastin Time (APTT) ≤ 1.5 ULN.
14. Women of childbearing potential should be ascetic or take contraception since the signing of ICF to 24 weeks or later after the last administration of drug.
15. Recovered from toxic effect of previous treatment (CTCAE ≤ 1), or related AE(s) is not defined as safety issue.
16. Catheter insertion is feasible and No White Blood Cells collection contraindications.

Exclusion Criteria:

1. Under pregnancy or lactation, or positive based on blood pregnancy test.
2. Severe allergic to related ingredients in the clinical trial.
3. Received any other investigational treatment within 4 weeks before the first administration or enrolled in another clinical trial the same time (exception: the other treatment is observational and non-investigational or the patient is under follow-up period)
4. Primary central nerve system (CNS) cancer, or subjects with CNS metastasis after localized treatment (except patients without CNS metastasis, clinically stable and neither steroid treatment nor treatment for CNS metastasis).
5. Patients with active autoimmune disease or require systemic steroid treatment. (except patients with cutaneous condition but without systemic treatment, or subjects with asthma in childhood but without intervention after grown-up, or subjects with hypothyroidism mediated by autoimmune dysfunction and receiving thyroxine as replaced treatment)
6. Immunodeficiency including HIV positive, harvested or natural immunodeficiency.
7. Patients with ≥ grade 3 thromboembolic events within 2 years or under thrombolysis treatment.
8. Patients with hereditary or acquired hemorrhagic disease
9. Patients with cardiovascular disease or symptoms:

   congestive heart failure (NYHA > 2); history of unstable angina pectoris; miocardial infarction within 48 weeks; clinically significant malignant arrhythmia (except atrial fibrillation and paroxysmal supraventricular tachycardia); Clinically significant prolonged QTcF (Male QTcF > 450 msec, Female QTcF > 470 msec); Uncontrolled hypertension.
10. Patients under active infection (except subjects with fever caused by tumor)
11. Patients with active tuberculosis, or history of active tuberculosis within 1 year before enrollment, or history of active tuberculosis over a year before enrollment but without standard treatment.
12. Patient with Active Hepatitis B or Active Hepatitis C.
13. Treponema pallidum antibody positive.
14. Received major surgery or under severe injury within 4 weeks before enrollment.
15. History of drug abuse, alcohol or drug addiction.
16. Received cell therapy before enrollment，such as TCR-T，CAR-T and TIL .
17. Allergic to IL-2.
18. Received treatment related chemo-therapy within 14 days of TC-E202 infusion (except lymphodepletion) .
19. Patient not suitable for the clinical trial according to investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity or Maximum Tolerated Dose (MTD) | Day 28 after the first TC-E202 infusion
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality recognized by SRC, and should be possibly related to TC-E202 cell therapy, and should be unrelated to the disease itself, disease progression, concomitant diseases or concomitant medication.
  The MTD is the highest dose at which ≤1 of 6 patients experienced a dose limiting toxicity (DLT) or the highest dose level studied if DLTs are not observed at any of the dose levels.
Overall response rate | Day0-Day730
  The efficacy of TC-E202 will be assessed by the objective response rate (ORR) is evaluated according to RECIST 1.1 and iRECIST. ORR is described as patients assessed with partial response (PR) and complete response (CR).
Treatment-related adverse events as assessed by CTCAE v5.0 | Day0-Day730
  The type, incidence and severity of adverse events include abnormal laboratory examination results with clinical significance after treatment, abnormal physical examination and blood examination results, bone marrow examination results, etc. Clinical and laboratory adverse events will be classified according to the National Cancer Institute general terminology standard for adverse events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Duration of response | Day0-Day730
  The efficacy of TC-E202 will be assessed by duration of response (DOR). The DOR refers to the length of time from the first appearance of a treatment response to the first occurrence of progressive disease or recurrence.
Progression free survival | Day0-Day730
  The efficacy of TC-E202 will be assessed by progression free survival (PFS). The PFS refers to the time from treatment to progressive disease or death for any reason.
Overall survival | Day0-Day730
  The efficacy of TC-E202 will be assessed by overall survival (OS). The OS refers to the time from treatment to death.
Maximum Persistence (Cmax) of TC-E202 | Day0-Day730
  Blood samples were collected to measure persistence of infused TC-E202 using polymerase chain reaction of a vector specific sequence in deoxyribonucleic acid (DNA) extracted from peripheral blood mononuclear cell (PBMC).
Time to Maximum Persistence | Day0-Day730
  Blood samples were collected to measure persistence of infused TC-E202 using polymerase chain reaction of a vector specific sequence in DNA extracted from PBMC.
Area Under the Plasma Concentration-time Curve From Zero to Day 28 (AUC[0-28]) | Day 28 after the first TC-E202 infusion
  Blood samples were collected to measure persistence of infused TC-E202 using polymerase chain reaction of a vector specific sequence in DNA extracted from PBMC.
Anti-PD-1 single chain antibody concentration | Day0-Day730
  The pharmacodynamics of TC-E202 will be assessed by Anti-PD-1 single chain antibody content.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoHua Wu, doctor, Study Director — Fudan University
Locations (1):
- Xiaochun Cheng, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No